CLINICAL TRIAL: NCT07152665
Title: The Effect of Video-Based Educational Content for Parents and Children on Anxiety, Fear, and Pain During Blood Draw in Children: A Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Murat Bektaş, Head of Department, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DokuzEU-5
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Pain; Fear Anxiety; Blood Drawing Procedure
Keywords: Children; Pain; Fear; Anxiety; Blood drawing procedure
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The population will consist of children between the ages of 4-7 who presented to Pediatric Phlebotomy Unit of the Central Laboratory at a university hospital in Turkey. The sample group will determined using stratified randomization based on strata created according to gender (female/male) and age (4, 5, 6, and 7 years). To calculate the required sample size, a repeated measures analysis of variance (ANOVA) was conducted using the G*Power software; the significance level was set at 0.01, statistical power at 99%, and a medium effect size was assumed. Based on these calculations, a minimum of 34 participants per group was required. Considering a potential 10% dropout rate, it was decided that each group would consist of 38 participants.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants in the study will assign using a stratified randomization method. Strata will create based on gender (two groups: female and male) and age (four groups: 4, 5, 6, and 7 years), and random sampling will perform within each stratum. The matching of the child with the nurse performing the blood draw will do randomly using the institution's routine queue management system. A nurse not involved in the study will assign each child to group and nurse who performing the blood draw based on their arrival number in the institution's blood draw queue system according to the previously determined randomization scheme. After the study is completed, the group names will be blinded, allowing analyses to be conducted without revealing the group names to the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimantel (Experimental): Parents of children in the intervention group will inform that the educational videos used in the study aim to reduce the child's pain, fear, and anxiety. An informational video willprepare by the researchers will show to the parents, while an age-appropriate video explaining the blood collection process will shown to the children.
  The video content wil structured in accordance with the existing literature Characters featured in the parent and child videos will select, and separate scenarios for each group will developed by the researchers. Video recordings will conduct outside of working hours in the blood collection unit, accompanied by a professional cameraman. To evaluate the feasibility and comprehensibility of the videos, a pilot study will conduct with five children and their parents who will not included in the main study.
  The parent video addressed the attitudes and behaviors that parents should exhibit before, during, and after the blood collection procedure.
  Interventions: Behavioral: Video-Based Education
- No Intervention: Control Group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Video-Based Education — Parents of children in the intervention group were informed that the educational videos used in the study aimed to reduce the child's pain, fear, and anxiety.
  Arms: Experimantel

SUMMARY:
This study aimed to examine the effect of video-based educational content prepared for parents and children on anxiety, fear, and pain levels experienced by children aged 4-7 during venipuncture procedures.

DETAILED DESCRIPTION:
This study aim to examine the effect of video-based educational content prepared for parents and children on anxiety, fear, and pain levels experienced by children aged 4-7 during venipuncture procedures.The study a single-centre, randomized controlled trial. The study will conduct in the pediatric phlebotomy unit of a university hospital's central laboratory in Turkey.

This randomized controlled trial will included 80 children aged 4-7, randomly assigned to intervention and control groups. The control group will receive routine clinical care before, during, and after venipuncture. In the intervention group, children and their parents will shown video-based educational content prior to the procedure. Data collection tools included a Child and Family Information Form, the Children's pain, Fear, and the Child Anxiety Scale. The normality of fear, anxiety, and pain scale scores will evaluate with the Shapiro-Wilk test. Repeated measures analysis of variance (ANOVA) will applied to compare scale scores across groups and time points. Within-group comparisons will conduct using one-way repeated measures ANOVA, while between-group differences at each time point were assessed with independent samples t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Children who will between the ages of 4-7,
* Children who will Blood collection procedure
* Have no cognitive development problems,

Exclusion Criteria:

* Children who will not want to participate in the study,
* Leave the research during the study,
* Have an audio-visual disorder that could prevent the use of video

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain Means | Five minutes before the blood draw attempt, during the blood draw attempt, and five minutes after the blood draw attempt
  Pain score will be measured with the Children's Pain Scale. The lowest score from the scale can be 0 and the highest score can be 10. As the score obtained from the scale increases, the child's pain increases. In this study, if children get high scores from the pianscale, it will be determined that they have high procedural pain. Getting a low score from the scale will indicate that their pain about the procedure is low.
Anxiety Means | Five minutes before the blood draw attempt, during the blood draw attempt, and five minutes after the blood draw attempt
  Anxiety score will be measured with the Child Fear and Anxiety Scale. The lowest score from the scale can be 0 and the highest score can be 10. As the score obtained from the scale increases, the child's anxiety increases. In this study, if children get high scores from the anxiety section of the scale, it will be determined that they have high procedural anxiety. Getting a low score from the scale will indicate that their anxiety about the procedure is low.
Fear Means | Five minutes before the blood draw attempt, during the blood draw attempt, and five minutes after the blood draw attempt
  Fear score will be measured with the Children's fear and anxiety scale. The lowest score from the scale can be 0 and the highest score can be 10. As the score obtained from the scale increases, the child's fear increases. In this study, if children score high on the fear section of the scale, it will be determined that their fear of the procedure is high. A low score on the scale will indicate that fears about the procedure are low.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Bektas, PhD, Principal Investigator — Dokuz Eylul University
Locations (1):
- School of Nursing, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, it is planned to be shared with other researchers after obtaining institutional permissions when they submit an application and provide their justification.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Andersson V, Bergman S, Henoch I, Simonsson H, Ahlberg K. Pain and pain management in children and adolescents receiving hospital care: a cross-sectional study from Sweden. BMC Pediatr. 2022 May 5;22(1):252. doi: 10.1186/s12887-022-03319-w. PMID 35513880
- [Background] Akkoyun S, Arslan FT, Sekmenli T. The effect of written document in perioperative information on the anxiety level and family-centered care of parents of children undergoing ambulatory surgery: A randomized controlled trial. J Pediatr Nurs. 2024 Mar-Apr;75:108-115. doi: 10.1016/j.pedn.2023.12.012. Epub 2023 Dec 25. PMID 38147711